CLINICAL TRIAL: NCT04172051
Title: The Effects of a Life Coaching Seminar on Gratitude and Psychological Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 121901
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Psychological; Depression, Anxiety; Psychological Stress; Mental Health Wellness 1; Mental Stress; Mental Depression
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Subjects will be admitted into the Tony Robbins event for free, or receive a voucher for an event in the future. The experimental group will attend the event. Subjects will be exposed to a variety of mind-body exercises and psychoeducational content including neural linguistic programming, designed to motivate, inspire, and improve the quality of people's lives. After attending the event, the experimental group will be asked to continue practicing "Priming " daily for a month. A One-page "priming" cheat sheet will be given to the subjects in the experimental group.
  Interventions: Behavioral: Tony Robbins Date with Destiny
- Control Group (No Intervention): The control group will be asked to engage in gratitude journaling every day for a month. The control group will NOT attend the event. This exercise will take 10 minutes to complete. The subject will write down three things that went well each day and provide an explanation about why they went well. This will be written down in a journal. The subjects will follow these instructions:
  1. Give the event a title (e.g., "co-worker complimented my work on a project")
  2. In the space below, write down exactly what happened in as much detail as possible, including what you did or said, and if other people were involved, what they did or said.
  3. Include how this event made you feel at the time and how this event made you feel later (including now, as you remember it).
- Motivated Experimental Group (Active Comparator): The Motivated Experimental Group (M Experimental) will consist of participants who registered and paid for Tony Robbins Date with Destiny (DWD). They are chosen as the motivated experimental as they will be paying full price for the event. The experimental group will attend the event. Subjects will be exposed to a variety of mind-body exercises and psychoeducational content including neural linguistic programming, designed to motivate, inspire, and improve the quality of people's lives. After attending the event, the experimental group will be asked to continue practicing "Priming " daily for a month. A One-page "priming" cheat sheet will be given to the subjects in the experimental group.
  Interventions: Behavioral: Tony Robbins Date with Destiny

INTERVENTIONS:
Behavioral: Tony Robbins Date with Destiny — DWD is a 6-day immersive transformational experience led by Tony Robbins. It will be held at the PALM BEACH, FLORIDA Convention Center from December 5th through December 10th. Subjects will be exposed to a variety of mind-body exercises and psychoeducational content including neural linguistic programming, designed to motivate, inspire, and improve the quality of people's lives.
  Arms: Experimental Group; Motivated Experimental Group

SUMMARY:
This study will consist of a randomized experimental group and a control group, In addition to the control and experimental group, there will also be a non-randomized motivated experimental group. Approximately 75 males and females from the ages of 18 to 80 will take part in this study. Subjects will be randomly divided into a Control and Experimental Group. Subjects for the control and experimental group will be recruited from a Tony Robbins Facebook page, and subjects in the experimental group (DWD Group) will be admitted to the Tony Robbins Date With Destiny Event (December 2019) in West Palm Beach for free, while the subjects randomly assigned to the control group, will not attend the event, but instead be required to a Gratitude Journaling experiment (Three Good Things Intervention). Psychological assessment surveys will be taken before the event, directly after the event, and one month following the event. The control group will take the psychological assessment before beginning journaling, directly after completing journaling, and one month following completion of journaling.

DETAILED DESCRIPTION:
Background:

A Pubmed or Google Scholar search reveals zero peer-reviewed articles examining Robbins' events, techniques, or principles, despite Robbins' enormous impact on culture, psychology, and individual lives. Furthermore, only poorly conceptualized studies testing clinically irrelevant hypotheses were ever conducted on Neurolinguistic Programming (NLP), a constitutive framework for part of Robbins' methodologies. Due to the intimate link between beliefs, wellness, and disease, the investigators hypothesize that an intervention focused on belief-restructuring, trauma release, psychoeducation, hope, inspiration, & social support like participation in a Tony Robbins' event (e.g. DWD) will demonstrate significant mental and physical health outcomes.

The investigators hope to obtain a better understanding of:

1. Whether Tony Robbins' DWD improves affect, depression symptoms, and well-being.
2. Setup collaboration infrastructure and generate hypotheses for a future randomized controlled trial to determine short- and long-term physiological and health effects of Tony Robbins' interventions.

Importance:

Tony Robbins, inventor of the term, life coach, and a coach to leaders around the world, regularly sells out 14,000 person arenas worldwide to talk about psychology, mental health, and wellbeing, and his website alone averages 1,000,000 unique visitors per month. Yet, a literature search through PubMed & Google Scholar reveals 0 empirical studies of Tony Robbins' work. Considering patients prefer psychotherapy over medication, there are a rich set of interventions to draw from Tony Robbins that could prove to be effective, accessible, and affordable in treating & preventing mental health issues including depression and suicide. Understanding the science of Tony Robbins' work could provide new theoretical frameworks and clinical interventions to inform non-pharmacological approaches to mental health.

Methodology:

This study will consist of a randomized experimental group and a control group, In addition to the control and experimental group, there will also be a non-randomized motivated experimental group. Approximately 75 males and females from the ages of 18 to 80 will take part in this study. Subjects will be randomly divided into a Control and Experimental Group. Subjects for the control and experimental group will be recruited from a Tony Robbins Facebook page, and subjects in the experimental group (DWD Group) will be admitted to the Tony Robbins Date With Destiny Event (December 2019) in West Palm Beach for free, while the subjects randomly assigned to the control group, will not attend the event, but instead be required to a Gratitude Journaling experiment (Three Good Things Intervention).

Subjects will be recruited by posting a Survey Monkey link on the DWD Facebook page as well as via email and direct referral. All participants will complete a consent form and take a brief eligibility survey administered digitally through Survey Monkey's secure system. Both groups will be given surveys before DWD, immediately after DWD to assess acute changes, and after 1 month after DWD to assess longitudinal changes. The experimental group will attend DWD. After attending DWD, the experimental group will be asked to continue practicing "Priming " daily for a month. A One-page "priming" cheat sheet will be given to the subjects in the experimental group. The control group will be asked to engage in gratitude journaling (protocol below) every day for a month. The control group will NOT attend the event.

A third group called the Motivated Experimental Group (M Experimental) will consist of participants who registered and paid for Tony Robbins Date with Destiny (DWD). They are chosen as the motivated experimental as they will be paying full price for the event. Subjects will be recruited at the event, as well as through the facebook group. Two investigators will follow up with subjects monthly by phone to assure consistency.

All surveys will be administered electronically through survey monkey. Informed Consent forms will also be provided electronically to all subjects. All subjects that participate in this study will receive a free book and audiobook, regardless of the group they were in upon completion of the study.

Study variables

Primary variables:

* Mental Health (depression, anxiety, stress) scores.

IRBs will need to be Electronically Signed by all participants. All Variables will be collected electronically over Survey Monkey. All questions will be extracted and worded directly off of the physical copy of each questionnaire into Survey Monkey.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18+, male and female, English speaking, lives in the U.S.
* Experimental group: must be a registered participant in Tony Robbins Palm Beach DWD (Dec 5th-10th)
* Control group: PHQ 9 score > 4 (5 is the cutoff for mild depression).

Exclusion Criteria:

* Excluded from the experimental group if you DO NOT attend the event.
* Excluded from the control group if you DO attend the event.
* Excluded from the Motivated Experimental Group if they have been compensated for their admissions fee.
* No confounding medical conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Changes in Patient Health Questionnaire - 9 (PHQ-9) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The PHQ-9 is a self-administered survey used for diagnosing depression and assessing depression severity. It measures each of the 9 Diagnostic and Statistical Manual of Mental Disorders-IV/V diagnostic criteria for depression on a 0-3 scale. Depression Severity is measured as follows: 0 none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against structured clinical interviews. PHQ-9 scores ≥10 exhibited a sensitivity of 88% and a specificity of 88% for major depression.
Date With Destiny Survey | Pre - Event
  Subjects will be asked if they have been to DWD or Not Been to DWD
Tony Robbins Events Survey | Pre - Event
  Subjects will be asked if they have been to any Tony Robbins events or not.
Tony Robbins Priming Techniques Survey | 1 Month Post - Event
  DWD subjects will be asked if they continued to use Tony Robbins Priming techniques daily for a month.
Changes in Generalize Anxiety Disorder - 7 (GAD-7) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The GAD-7 is a self report-based survey that assesses generalized anxiety disorder and severity on a 7-item scale. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. The GAD-7 was compared to diagnoses by mental health professionals. Using scores >/= 10, It has sensitivity of 89% and specificity of 82%.
Changes in Perceived Stress Scale (PSS-10) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Perceived Stress Scale-10 (PSS-10) measures global perceived stress via self-report on a ten item scale. Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Total scores ranging from 0-13 would be considered low stress. Total scores ranging from 14-26 would be considered moderate stress. Total scores ranging from 27-40 would be considered high perceived stress.
Changes in PERMA Profiler | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The scale measures five aspects of well-being defined by Martin Seligman, PERMA - positive emotion, engagement, relationships, meaning, and accomplishment, as well as negative emotion and health.
Changes in Dysfunctional Attitudes Scale - 17 (DAS-17) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Attitudes Scale-17 is a short form version of the DAS-A rated on a 7-point Likert scale (7 = fully agree; 1 = fully disagree). It is comprised of two subscales, perfectionism (11-77) and dependency (6-35), as well as a total score (17-119). Higher scores indicate higher levels of dysfunctional attitudes.
Changes in Primals Inventory -18 (PI-18) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Primal World Beliefs Index-18 is a short form version of the PI-99 that measures beliefs about the world in general through four constructs, Safe, Enticing, and Alive, and the overall construct, Good. Each construct is on a scale of 0-5, with higher scores indicating higher levels of Good, Safe, Enticing, and Alive.
Changes in Satisfaction with Life Survey | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Satisfaction with life scale is a five question survey scored on a 7-point Likert scale with scores ranging from 5-35, with 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied. The coefficient alpha for the scale has ranged from .79 to .89, indicating that the scale has high internal consistency. The scale was also found to have good test-retest correlations (.84, .80 over a month interval).
Changes in Close Relationships Questionnaire | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Close Relationships Questionnaire is a 36 question survey that measures attachment anxiety and attachment avoidance. It is scored on a Likert scale from 1 to 7 with total scores ranging from 36 to 252.
Changes in Sexual Satisfaction | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The sexual satisfaction scale is a 4 question scale on a six point Likert scale ranging from extremely dissatisfied to extremely satisfied, with scores ranging from 4 to 24. Higher scores indicate higher sexual satisfaction. The scale is a brief assessment of sexual satisfaction and shouldn't be used for studies focused on sexuality.
Changes in Adult Hope Scale | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Adult Hope Scale is a 12 item scale on an 8 point Likert scale ranging from definitely false to definitely true with scores ranging from 12 to 96. Higher scores indicate a higher positive motivational state. The scale seeks to measure hope in terms of motivation.
Changes in Gratitude Questionnaire | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Gratitude Questionnaire is a 6 item questionnaire scored on a 7 point Likert scale ranging from strongly disagree to strongly agree with scores ranging from 6 to 42. Higher scores indicate more gratitude experienced in daily life. The scale seeks to measure differences in proneness to experience gratitude in daily life.
Changes in Adverse Childhood Experience (ACE) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  The Adverse Childhood Experiences questionnaire is a ten question survey assessing incidence of common traumas before age 18. Scores range from 0-10, with higher scores indicating higher levels of childhood trauma.
Changes in Date With Destiny - Specific Surveys | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  Date With Destiny - Specific Surveys will be used to assess specific and measurable before and after psychometric, health, and lifestyle changes.
Changes in Short Form Survey-36 (SF-36) | Pre - Event, 24 hours Post - Event, 1 Month Post - Event
  Health Status Questionnaire will be used to assess changes in health before and after the event.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University Department of Genetics, Stanford, California
  - The Applied Science and Performance Institute, Tampa, Florida
  - Palm Beach County Convention Center, West Palm Beach, Florida

IPD SHARING:
Plan to Share IPD: No